CLINICAL TRIAL: NCT05471700
Title: To Evaluate Safety and Efficacy of Azacitidine Combination With Venetoclax for Treatment of Newly Diagnosed Fit Acute Myeloid Leukemia Patients：A Multicenter, Single-arm Study
Brief Title: Single Arm Study of Azacitidine and Venetoclax for Treatment of Newly Diagnosed Fit Acute Myeloid Leukemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA+Venetoclax
Record Dates: First submitted 2022-07-01; First posted 2022-07-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; Newly Diagnosed AML; Azacitidine; Venetoclax; Induction Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine combined with Venetoclax (Experimental): Each course is 28 days long. Subjects with newly diagnosed AML receive Venetoclax once daily by oral. The doses of Venetoclax is 100 mg on Day 1, 200 mg on Day 2, reaching a target dose of 400 mg on Day 3 and continuing through Day 28. If concomitantly receiving azoles, the dose of Venetoclax will be adjusted according to the instructions. At the same time patients will receive Azacitidine 75mg/m2 subcutaneous on Days 1-7.The induction therapy includes 1-2 cycle until subjects get remission.
  Once complete remission, subjects will receive consolidation. Azacitidine combined with Venetoclax or middle to high dose of arabinoside based chemotherapy would be given at the discretion of the physician.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Subjects will receive Azacitidine 75 mg/m2 on days 1-7.Each course is 28 days long.
  Other Names: 5-Azacitidine; 5-aza
Drug: Venetoclax — Subjects would receive Venetoclax once daily by oral. The doses of Venetoclax is 100 mg on Day 1, 200 mg on Day 2, reaching a target dose of 400 mg on Day 3 and continuing through Day 28. Each course is 28 days long.
  Other Names: Venclexta; Venclyxto

SUMMARY:
The goal of this clinical research study is to evaluate the safety and efficacy of Azacytidine in combination with Venetoclax in patients with newly diagnosed fit acute myeloid leukemia.

DETAILED DESCRIPTION:
The Study Drug:

Azacitidine is a DNA Demethylated drug, which is approvd for treatment of elderly AML patients Venetoclax targets the anti-apoptotic protein Bcl-2 and the process of oxidative phosphorylation to induce apoptosis of leukemia cells and exhibits anti-tumor activity.

Study Group:

single arm: AZA plus Venetoclax

Study Drug Administration:

Each course is 28 days long. Venetoclax is taken once daily by oral. The doses of Venetoclax is 100 mg on Day 1, 200 mg on Day 2, reaching a target dose of 400 mg on Day 3 and continuing through Day 28. If concomitantly receiving azoles, the dose of Venetoclax will be adjusted according to the instructions. Azacitidine is taken 75mg/m2 on Days 1-7. Subjects would received 1-2 cycles induction therapy. Once get remission, subjects would received the same indution therapy of middle to high dose of cytarabine based chemotherapy at the discretion of the physician for consolidation. Allo-HSCT is suggested for subjects with the moderate to adverse ELN2017 risk.

Study Visit:

After treatment, relapse and survival will be followed monthly by telephone, on-site visits, and/or study medical records for up to two years (calculated from the first day of induction therapy); Thereafter follow-up every 3 months for one year.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 45 to 65 years old,both male and female
* 2.Be able to understand and sign informed consent
* 3.Untreated AML patients (non-APL) diagnosed according to the 2016 World Health Organization (WHO) classification and diagnostic criteria for acute myeloid leukemia
* 4.Patients with an ECOG performance status 0,1,2 or 3
* 5.Expected survival time≥3 months
* 6.Laboratory indicators meet the following standards:

  1. Bilrubin, ALT and AST were all less than 3 times the upper limit of normal within 7 days before the first day of treatment
  2. Serum creatinine clearance rate is greater than 30ml/min

Exclusion Criteria:

* 1.patients participating in other interventional or observational clinical studies currently
* 2.Patients has a history of myeloproliferative neoplasm [MPN]
* 3.Patients with acute promyelocytic leukemia
* 4.Active CNS involvement in patients with acute myeloid leukemia
* 5.Patients with active hepatitis B or C, HIV infection before enrollment
* 6.Cardiovascular status of patients evaluate by NYHA classification method > 2
* 7.Patients have chronic respiratory disease requiring continuous oxygen treatment, or any sitiuation investigator believes will adversely affect this study (including renal, neurological, psychiatric, endocrine, metabolic, immune, hepatic, cardiovascular disease and known history of allergy to any study drug)
* 8.Patients suffering from malabsorption syndrome or other diseases that prevent the enteral route of administration
* 9.patients present with an uncontrolled systemic infection (viral, bacterial, or fungal)
* 10.Patients with a history of other malignancies within 2 years before enrollment, except for the following cases:

  1. Adequately treated carcinoma in situ of the cervix or carcinoma of the breast
  2. Basal cell carcinoma or localized squamous cell carcinoma of skin

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 36 months
  ORR is defined as the percentage of participants who achieve the CR + CRi + Partial Remission (PR) as evaluated by the investigator.

SECONDARY OUTCOMES:
Minimal residual disease (MRD) negative response rate | Up to 36 months
  The number of subjects who obtained MRD negative as a percentage of all evaluable subjects.
Duration of Remission (DOR) | Up to 36 months
  From the first achievement of PR, CR, or CRi to time of disease progression
Allogeneic Hematopoietic Stem Cell Transplantation Rate | Up to 36 months
  Proportion of subsequent allogeneic hematopoietic stem cell transplantation in intermediate-risk and adverse-risk patients
Overall Survival (OS) | Up to 36 months
  From start of protocol treatment to time of death due to any cause, or until last follow-up
Event-Free Survival (EFS) | Up to 36 months
  From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier; or until last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yuhua Li, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Nanfang Hospital of Southern Medical University, Guanzhou, Guandong, China

IPD SHARING:
Plan to Share IPD: Yes
We will share our data within 6 months after the end of the trial. You can ask us for data or obtain it on the Clinical Trial Management Public Platfcrm of clinical trial.
  Supporting Information: Study Protocol
Supporting Information: Study Protocol
Time Frame: The data will be available and permanently disclosed within 6 months after the trial.
Access Criteria: You can log in to the website for data access or contact us for data.